CLINICAL TRIAL: NCT02063074
Title: Bone, Endocrine and Lifestyle Longitudinal Study
Acronym: BELLS
Status: Terminated | Type: Observational
Why Stopped: Lack of participants and funding support
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, Assistant Professor, University of Southern California
Other Study IDs: HS-13-00789
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be tested for lipids, glucose, insulin, estrogens, bone biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this proposal is to determine the long-terms effects of hormone and lifestyle factors on bone health in young women over a 20-year time period. It is our primary hypothesis that premenopausal women with irregular periods or endocrine issues related to estrogen will have significantly poorer low back and hip bone health when compared to regularly menstruating women. It is our secondary hypothesis that long-term assessment of changes in endocrine function and lifestyle behaviors will assist in establishing risk factors for osteoporosis in young women. This study will include 1000 premenopausal women. The women will participate in the collection of a blood sample, bone scan, body fat measures, and lifestyle questionnaires. In addition, we hope to use this initial study to develop a group of women to follow throughout menopause, with additional visits occurring every 5 years over the course of their life.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age
* free from any uncontrolled chronic disease that may affect bone mass
* Not pregnant

Exclusion Criteria:

* Women recently diagnosed with uncontrolled chronic disease(s) at time of enrollment known to affect bone mass, including but not limited to metabolic and endocrine diseases (specifically, diseases of the thyroid and parathyroid glands), osteoporosis, and those women who have taken prophylactic bone density agents, such as Fosamax.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Premenopausal women over the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Principal Investigator — University of Southern California
Locations (1):
- Women's Health and Exercise Laboratory, University of southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided